CLINICAL TRIAL: NCT06213740
Title: Validation of a New Simplified Scoring System (ACME) for Acute Calculous Cholecystitis
Brief Title: Validation of a New Simplified Scoring System for Acute Calculous Cholecystitis
Acronym: ACME
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: ACME_Validation
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Acute Cholecystitis
Keywords: Acute Cholecystitis; Cholecystectomy; Tokyo Guidelines; Postoperative Complications; Mortality; High-risk patient
MeSH Terms: conditions — Cholecystitis, Acute; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute calculous cholecystitis (ACC) is the second most frequent surgical condition in emergency departments. The recommended treatment is surgical treatment (ST) and the accepted mortality is <1%, but in severe and/or fragile patients is higher. Despite the Tokyo Guidelines, there no consensus on who is the unfit patient for ST. A recent study has identified 4 risk factors that predicts the mortality in a 92% of patients (ACME) and could help to develop new guidelines in ACC. The aim of this study is this validation of the new simplified scoring system for mortality in ACC.

DETAILED DESCRIPTION:
This is a retrospective single-center observational study of 387 adults with ACC during 2 non-consecutive years (2017/2021), including baseline demographic characteristics, comorbidity severity defined as Charlson Comorbidity Index (CCI), ASA Score, Tokyo Guidelines' severity classification and the new ACME Score. The primary outcome is to study the prediction of mortality of ACME score. Secondary outcomes include complications following Clavien-Dindo's classification, C-statistic, and ROC Curves.

ELIGIBILITY:
Inclusion Criteria:

* The selected patients were among those who had acute cholecystitis according to the TG18 or received a diagnosis of ACC in the histopathological report.

Exclusion Criteria:

* The study case definition was a "Pure ACC", therefore, patients with any other concomitant diagnosis potentially influencing outcome such as acute pancreatitis, acalculous cholecystitis, chronic cholecystitis, acute cholangitis, postoperative cholecystitis, gallbladder adenocarcinoma and those who had undergone cholecystectomy as a prophylactic measure in another intervention were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the admisions with the inclusion criteria during 2017 and 2021.
Sampling Method: Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Mortality | 2017 and 2021
  Evaluate the mortality in the cohort

SECONDARY OUTCOMES:
Complications | 2017 and 2021
  Clavien-Dindo

CONTACTS AND LOCATIONS:
Locations (1):
- Ana María González Castillo, Cerdanyola del Vallès, Barcelona, Spain